CLINICAL TRIAL: NCT01784666
Title: Adjunctive Isradipine for the Treatment of Bipolar Depression
Acronym: Isradipine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Roy Perlis, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-P-002449/1
Record Dates: First submitted 2013-02-04; First posted 2013-02-06 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Depression; Lithium; Valproate; Isradipine
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Isradipine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Isradipine-Isradipine (Experimental): Subjects will receive isradipine in phase 1 (4 weeks) and phase 2 (4 weeks)
  Interventions: Drug: Isradipine
- Placebo -> Isradipine (Experimental): Placebo non-responders after the 1st 4 weeks will be re-randomized 1:1 to placebo or isradipine for the next 4 weeks
  Interventions: Drug: Isradipine; Drug: Placebo
- Placebo-Placebo (Placebo Comparator): Placebo nonresponders for the 1st 4 weeks will be re-randomized 1:1 to placebo or isradipine for the subsequent 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Isradipine — The study uses the Sequential Parallel Comparison design (SPCD), with two 4-week phases: n=30 subjects are randomized 1:1 to isradipine versus placebo add-on for 4 weeks, with the placebo nonresponders re-randomized 1:1 for a further 4 weeks. The SPCD will allow us to pool data from both phases to estimate the isradipine treatment effect. Subjects who respond in phase 1, and all subjects who receive isradipine in phase 1, continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed.
  Arms: Isradipine-Isradipine; Placebo -> Isradipine
Drug: Placebo — Subjects (n=15) are randomized to placebo add-on for 4 weeks, with the nonresponders re-randomized 1:1 to isradipine vs placebo for a further 4 weeks. Subjects who respond in phase 1 continue blinded treatment in phase 2 to preserve the blind, but only phase 1 results are analyzed.
  Arms: Placebo -> Isradipine; Placebo-Placebo

SUMMARY:
This study investigates the medication isradipine, which is currently approved by the FDA to treat high blood pressure, in the treatment of depression in bipolar disorder. Isradipine or placebo (contains no active medication) will be used as an "add-on" to lithium, valproate, and/or atypical antipsychotics for individuals currently experiencing a major depressive episode. Our hypothesis is that isradipine will be superior to placebo in improving depressive symptoms.

DETAILED DESCRIPTION:
Primary Aim: To estimate the antidepressant efficacy of isradipine versus placebo as an adjunct to lithium, valproate, and/or other atypical antipsychotics among individuals with bipolar I disorder in a nonpsychotic major depressive episode.

Hypothesis: Isradipine will be superior to placebo in improvement of depressive symptoms assessed by the Montgomery-Asberg Depression Rating Scale (MADRS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* written informed consent
* meets Diagnostic and Statistical Manual-IV (DSM-IV) criteria (by Structured Clinical Interview for Diagnostic and Statistical Manual - IV -I/P (SCID)) for bipolar I disorder, current episode depressed
* Montgomery-Asberg Depression Scale (MADRS) score of at least 20 (i.e., moderate depression) and no greater than 34 (i.e., severe depression) at screen and baseline visit
* Young Mania Rating Scale (YMRS) score < 12 at screen and baseline visit
* currently treated with a lithium preparation (carbonate or citrate) at stable dose for at least 4 wks with level >0.6 and <1.0; and/or valproate at stable dose for at least 4 wks at level >60 and <110; and/or other atypical antipsychotic at stable dose for at least 4 weeks (at least minimum FDA-labeled dose)
* Caucasian by self-report - please see discussion below

Exclusion Criteria:

* Psychotic features in the current episode, as assessed by YMRS item #8 > 6 [where treatment guidelines urge use of antipsychotics that may confound isradipine results]
* felt by the study clinician to require inpatient hospitalization for adequate management (to include serious suicide or homicide risk, as assessed by evaluating clinician)
* 3 or more failed pharmacologic interventions in the current major depressive episode, excluding lithium/valproate/other atypical antipsychotic [response rates for these subjects is likely to be extremely low and would require a substantially larger-scale study to identify treatment effects]
* obsessive-compulsive disorder, or any diagnosis of a DSM-IV anxiety disorder where the anxiety disorder and not bipolar disorder is the primary focus of clinical attention
* current substance use disorder other than nicotine, by SCID-I/P
* a primary clinical diagnosis of a personality disorder, or comorbid diagnosis of antisocial or borderline personality disorder
* pregnant women or women of child bearing potential who are not using a medically accepted means of contraception (to include oral contraceptive or implant, condom, diaphragm, spermicide, intrauterine device, tubal ligation, or partner with vasectomy)
* women who are breastfeeding
* other unstable medical illness including cardiovascular, hepatic, renal, respiratory, endocrine, neurological, or hematological disease, based on review of medical history, physical examination, and screening laboratory tests (this will include any clinical or laboratory evidence of hypothyroidism; if maintained on thyroid medication must be euthyroid for at least 1 month before Visit 1)
* history of hypertension or current treatment for hypertension
* current use of isradipine or history of anaphylactic reaction or intolerance to isradipine or any component of the preparation
* ECG abnormalities at entry: prolonged QTC interval or complete or incomplete bundle branch block
* patients who have taken an investigational psychotropic drug within the last 3 months
* patients receiving other excluded antipsychotics or antidepressants within 2 weeks prior to study entry
* patients requiring continued treatment with excluded medications (see below).

Excluded medications: antidepressants, antipsychotics, and anticonvulsants (other than valproate), which could influence calcium signaling or impact mood; other calcium channel blockers; any other antihypertensive because of the risk of cause hypotension; any other drug known to interact with isradipine. Benzodiazepines or other sedative-hypnotic agents (e.g., zolpidem) may not be initiated after study entry; subjects requiring these agents will be removed from the study. Allowed: Sedative-hypnotic agents if dosage has been stable for 4 weeks prior to study entry; thyroid or estrogen replacement provided dosage has been stable for 3 months. Acceptable anticonvulsants include lamotrigine, valproate, gabapentin, topiramate, oxcarbazepine, carbamazepine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy H Perlis, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Isradipine-Isradipine | Placebo -> Isradipine | Placebo-Placebo
Started | 1 | 0 | 1
Completed | 1 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Isradipine-Isradipine | Placebo -> Isradipine | Placebo-Placebo | Total
Number analyzed (Participants) | 1 | 0 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 56 [56 to 56] |  | 44 [44 to 44] | 50 [44 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS (4 Weeks)
Description: Change in Montgomery-Asberg Depression Rating Scale (MADRS) in isradipine-treated epochs versus placebo-treated epochs.
  These scores represent total scores, and on the MADRS total scores range from 0-60. A higher score indicates increased depression severity.
Time Frame: Baseline vs week 4 (and, for placebo nonresponders in 1st 4 weeks, week 8 vs week 4)
Measure: Number; unit: scores on a scale
Arm/Group | Isradipine-Isradipine | Placebo -> Isradipine | Placebo-Placebo
Number analyzed (Participants) | 1 | 0 | 1
scores on a scale | -9 |  | 0

ADVERSE EVENTS:
Arm/Group | Isradipine-Isradipine | Placebo -> Isradipine | Placebo-Placebo
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
The study was terminated early by the investigator because delays in study initiation and insufficient recruitment. Our statisticians have advised that this analysis is uninformative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No